CLINICAL TRIAL: NCT03707197
Title: The Impact of 8 Weeks of a Digital Meditation Application on Stress-Induced Eating
Brief Title: Guided Meditation and Stress-Induced Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: The University of California's Healthy Campus Network (Other); Headspace Meditation Limited (Industry)
Responsible Party: Principal Investigator, A. Janet Tomiyama, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Meditation and Eating
Record Dates: First submitted 2018-10-09; First posted 2018-10-16 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Stress-induced Eating
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Randomization to either digital meditation condition or waitlist-control condition
Who Masked: Investigator
Masking Description: Investigator will be blind to condition throughout data accrual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation Group (Experimental): The intervention group will be assigned to a digitally-based meditation intervention (Headspace app- Basic + Stress packs) and asked to use this for at least 10 minutes a day over the course of 8 weeks
  Interventions: Behavioral: Meditation
- Wait-list Control Group (No Intervention): Wait-list control group participants will continue their normal activities and not engage in any form of meditation during the study period

INTERVENTIONS:
Behavioral: Meditation — Ten minutes of meditation per day for 8 weeks using a mobile application
  Arms: Meditation Group

SUMMARY:
The aim of this study is to test the effects of a digital meditation intervention in a sample of UCLA employees who report mild to moderate stress. We will randomize University of California Los Angeles employees to either 8-weeks of a digital meditation intervention (using the commercially available application Headspace) or a waitlist control condition.

DETAILED DESCRIPTION:
The aim of this study is to test the effects of a digital meditation intervention in a sample of UCLA employees who report mild to moderate stress. UCLA employees will be randomized to either 8-weeks of a digital meditation intervention (using the commercially available application Headspace) or a waitlist control condition.

Participants who are assigned to the intervention group will be asked to download and use the Headspace mobile application for at least 10 minutes per day for 8 weeks. All participants will be asked to fill out short (no longer than 25 minutes) questionnaires at baseline, week 4, week 8 (post intervention), and a 4-month follow up period. Among participants who are randomized to the digital meditation intervention, they will also take part in a 1-year follow up. All activities will take place online (via computer or smartphone).

Prior to randomization, participants will complete an eligibility screening and complete the baseline questionnaire battery. The entirety of the study is digital and there are no in-person assessments. Adherence will be tracked remotely. The goal is to recruit as many as 1000 participants (500 per condition).

ELIGIBILITY:
Inclusion Criteria:

* Have access to a smartphone or computer everyday
* Are fluent in English
* Are a University of California, Los Angeles employee
* Report mild to moderate levels of stress
* Consent: demonstrate understanding of the study and willingness to participate as evidenced by voluntary informed consent and has received a signed and dated copy of the informed consent
* Are at least 18 years of age

Exclusion Criteria:

* You may not join if you are an experienced meditator or have participated in a formal meditation practice in the last 6 months (defined as once or more per week for a duration of 20 minutes or more at each practice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 943 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Reductions in perceived stress as measured by the Perceived Stress Scale | Baseline to post-intervention (8 weeks from baseline)
  Changes in the Perceived Stress Scale (range: 1-40; Cohen, Kamarck, & Mermelstein, 1988). Higher scores indicate greater psychological distress.

SECONDARY OUTCOMES:
Reductions in stress-induced eating as measured by the Palatable Eating Motives Scale | Baseline to post-intervention (8 weeks from baseline)
  Changes self-reporting using highly palatable foods to cope with stress, according to the Palatable Eating Motives Scale Coping subscale (range: 1-20) Burgess, Turan, Lokken, Morse, & Boggiano, 2014). Higher scores indicate a higher likelihood of using palatable foods to cope with stress.
Reductions in reward-based eating as measured by the Reward-based Eating Drive | Baseline to post-intervention (8 weeks from baseline)
  Changes in self-reporting intrinsic rewards from consuming highly palatable foods, according to the Reward-based Eating Drive (RED) Scale (range: 1-45; Epel, et al. 2014). Higher scores indicate a greater reward response from consuming palatable foods.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Tomiyama, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided